CLINICAL TRIAL: NCT02303834
Title: Single Blinded Randomised Control Trial of Treatment of Sleep Disordered Breathing in Preeclampsia With Nasal CPAP
Brief Title: CPAP in Preeclampsia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Sydney (Other)
Collaborators: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Principal Investigator, Professor David Celermajer, Professor, University of Sydney
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC 14/092
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Preeclampsia; Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): The control group will not be fitted with CPAP.
- CPAP group (Experimental): The group will wear a CPAP device throughout the night. The mask fits comfortably over the nose and delivers a steady stream of air under slight pressure (auto-set).
  Interventions: Device: Continuous Positive Airway Pressure Ventilation (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure Ventilation (CPAP) — A mask worn over the nose that delivers air under slight pressure.
  Arms: CPAP group

SUMMARY:
Study design:

Single blinded randomised control trial

Planned sample size:

30 (women randomized 2:1 to receive either CPAP or no CPAP)

Objectives:

Primary objective: Assess the effects of nasal CPAP on sleep physiology, 24 blood pressures and fetal movements in pregnant women (24-37 weeks gestation) with preeclampsia.

Secondary objective: Assess baseline sleep physiology, blood pressure control and fetal well-being in pregnant women (24-37 weeks gestation) with preeclampsia by completing sleep studies, 24 hour blood pressure monitors, CO2 monitors, and nocturnal fetal movement and HR monitors.

Study Procedure:

Participants will be recruited from the antenatal ward or high-risk antenatal clinic. Following informed consent participants will be randomly assigned to receive either CPAP or no CPAP for one night, following an initial baseline overnight sleep study.

Baseline- Night 1

1. Sleep study with fetal movement and HR monitor
2. 24 hour BP monitor
3. CO2 monitor

Intervention- Night 2 (Nasal CPAP device or no CPAP)

1. Sleep study with fetal movement and HR monitor
2. 24 hour BP monitor
3. CO2 monitor

Post-partum questionnaire A brief questionnaire to be completed within the first 6 weeks post-partum related to the participant's personal health, their child's birth details and health.

DETAILED DESCRIPTION:
DESIGN Single blinded randomized control trial STUDY GROUPS Women diagnosed with preeclampsia by their treating physicians (BP>140/90 and proteinuria> 300mg in 24 hours) who are being managed either as inpatients or out-patients. They will be randomized in a 2:1 ratio to receive active CPAP or no CPAP either in hospital (if they are inpatients) or at home (outpatients).

NUMBER OF PARTICIPANTS A total of 30 women will be recruited. NUMBER OF CENTRES This study will be conducted at 2 centres- Royal Hospital for Women, Randwick and Royal Prince Alfred Hospital, Camperdown. The aim will be to recruit 15 participants from each site.

INTERVENTIONS The intervention is nasal CPAP. The intervention group will be fitted with nasal CPAP on night 2, set to deliver positive pressure airway ventilation. The control group will not receive CPAP on night 2. The CPAP devices to be used are the ResMed S9 and the Philips Respironics REMstar Pro, both of which are automatically setting machines that respond to the presence of snoring, partial airway obstruction and complete apneas and increase airway pressure to a therapeutic level. These systems are commercially available and in widespread everyday routine clinical use in Australia. Nasal CPAP has been used for over 30 years including in pregnant women and has been found to be very safe therapy.

DURATION Participants will be required to undertake 2 overnight sleep studies/BP monitors/CO2 monitors and complete a 10 minute questionnaire in the first 6 weeks post-partum. The study will be undertaken between 1/6/14 to 1/6/16.

INVESTIGATION PLAN Following informed consent participants will be enrolled to undergo the following investigational plan.

Baseline demographic data: all enrolled participants will be asked to provide the following information:

* age,
* gestation
* height
* current weight and pre-pregnancy weight
* medical history
* medications
* family history
* snoring history
* smoking and illicit drug taking history

They will then be asked to complete a Modified Epworth Sleepiness Scale questionnaire.

Overnight Sleep Study/ BP monitor and Fetal Monitor:

Inpatients will undertake a Sleep Study with accompanying 24 BP monitor, CO2 monitor and fetal movement/HR monitor in their hospital bed on the day of recruitment. Outpatients will be given the equipment and a brief lesson on its use by investigators on the day of recruitment, and asked to perform the study in their own homes. They will be asked to then return the equipment to the hospital the following day for analysis.

Second Night- Intervention On the subsequent day, the active group will be fitted with a nasal CPAP device and given a brief lesson on its use (Intervention group- CPAP, Controls- no CPAP). Inpatients will then complete a Sleep study, 24 hour BP monitor, CO2 monitor and fetal movements/HR monitor whilst on nasal CPAP. Outpatients will complete the same tests with nasal CPAP in their own homes. Outpatients will then return the equipment to the hospital for analysis the following day.

Sleep Study- Sonomat HST The Sonomat is a portable mat that is placed on top of the participant's mattress (underneath the sheets). It contains a microphone and four vibration sensors to detect breath sounds, breathing movements and body movement. It will assess snoring, the number of apneas, the number of hypopneas, the number of arousals, and hourly blood oxygen saturation (%) throughout the night. It also measures the total number of fetal movements throughout the night, and will be used to calculate average hourly fetal movements.

The Sonomat HST (ARTG number: Sleep Assessment Device 179807, software 179908) is registered with the Therapeutic Goods Administration and is routine use to perform ambulatory sleep assessments.

24 Hour BP monitor and CO2 monitor A blood pressure cuff will be applied to the left upper arm for 24 hours. It will inflate hourly to measure the participant's systolic and diastolic blood pressure (mmHg) and will record all values. From this average nocturnal and daytime BPs will be calculated. The device to be used is a Spacelabs portable oscillometric system ABP 20217.

The CO2 monitor is a transcutaneous monitor applied to the patient's earlobe which continuously measures CO2, O2 and HR. From this, we can monitor alterations in CO2 and O2 such as desaturations, complete apnoeas and hypercapnic episodes.

Nasal CPAP (Continuous positive airway pressure) The CPAP devices used are ResMed S9 or Philips-Respironics REMstar Pro, which are automatically setting machines that respond to the presence of upper airway obstruction and complete apneas and increase airway pressure to a therapeutic level.

The CPAP system is a small machine that sits at the bedside with a mask attached to the machine via a tube. The mask fits comfortably over the nose and delivers a steady stream of air under slight pressure (auto-set). It is to be worn throughout the night whilst the participant sleeps. Modern nasal CPAP masks and nasal pillow are very comfortable, and provided there is a gentle background flow of air, they are very easy to use and allow normal sleep.

Post-partum questionnaire All participants will be asked to complete a brief questionnaire, which will be sent to them via email or conventional mail, in the first 6 weeks post-partum. This will ask questions regarding their gestation at delivery, fetal birth weight, maternal and fetal health and current signs/symptoms of sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* Women 24-37 weeks pregnant
* Singleton pregnancy
* Primiparous and primigravid
* Maternal age 18-45 years
* Diagnosis of preeclampsia by their treating specialist (SBP>140/90 and proteinuria>300mg in 24 hours)

Exclusion Criteria:

* A previous diagnosis of hypertension, cardiac, respiratory or renal disease.
* Any regular cardiac or respiratory medications (PRIOR to pregnancy and diagnosis of preeclampsia)
* Current smokers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maternal Blood Pressure | 2 days
  Maternal blood pressure will be measured hourly for 48 hours during the 2 days of the study. This will be used to compare average nocturnal and daytime blood pressures between the first and 2nd (intervention) night in the 2 groups.
Fetal movements | 2 days
  Fetal movements will be measured throughout the night for 2 consecutive nights (night 1 and night 2-intervention). This will be used to calculate average fetal movements per hour in each of the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Sullivan, MBBS phD, Study Chair — University of Sydney
Locations (2):
- Australia (2):
  - Royal Hospital for Women, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No
Data is de-identified and analysed as a cohort, no individual data will be published.